CLINICAL TRIAL: NCT03798782
Title: Ross for Valve Replacement in AduLts Trial
Acronym: REVIVAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Richard Whitlock, Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REVIVAL-2018
Record Dates: First submitted 2018-12-18; First posted 2019-01-10 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Aortic Valve Disease
Keywords: Cardiac surgery; Aortic valve replacement; Ross procedure
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ross procedure (Experimental): The patient will undergo the Ross procedure where the surgeon will replace the aortic valve using a pulmonary autograft (Ross procedure) with pulmonary homograft replacement of the pulmonary root.
  Interventions: Procedure: Ross procedure
- Conventional aortic valve replacement (Active Comparator): The patient will undergo Conventional aortic valve replacement where the surgeon will replace the aortic valve with another prosthesis which can include a mechanical prosthesis, a stented biological prosthesis, a stentless biological valve or root, or a catheter valve.
  Interventions: Procedure: Conventional aortic valve replacement

INTERVENTIONS:
Procedure: Ross procedure — The patient will undergo the Ross procedure where the surgeon will replace the aortic valve using a pulmonary autograft (Ross procedure) with pulmonary homograft replacement of the pulmonary root. Identified Ross experts will perform all Ross procedures.
  Arms: Ross procedure
Procedure: Conventional aortic valve replacement — The patient will undergo Conventional aortic valve replacement where the surgeon will replace the aortic valve with another prosthesis which can include a mechanical prosthesis, a stented biological prosthesis, a stentless biological valve or root, or a catheter valve.
  Arms: Conventional aortic valve replacement

SUMMARY:
This study evaluates two methods of aortic heart valve replacement in adults aged 18-60, the Ross procedure versus conventional aortic valve replacement using a biologic or mechanical heart valve. The Ross procedure replaces a patient's diseased aortic valve with his/her own pulmonary valve and uses a donor valve in the pulmonary position which receives less stress than the aortic valve. Mechanical valves tend to form blood clots so they need long-term blood thinners that increase risk of bleeding and lower quality of life. Animal tissue valves reduce clotting and bleeding risks but wear out sooner and shorten patient life-span.

DETAILED DESCRIPTION:
Heart valves help control blood flow through the heart and, if diseased, may need to be replaced. After having a heart valve replaced, patients have a higher risk of death than people who have not had a valve replaced. In young adult patients, replacing the aortic heart valve with a mechanical valve halves their life-span compared to other people their age. Mechanical valves tend to form blood clots so they need long-term blood thinners that increase risk of bleeding and lower quality of life. Animal tissue valves reduce clotting and bleeding risks but wear out sooner and shorten patient life-span. An operation, called the Ross procedure, replaces a patient's diseased aortic valve with his/her own pulmonary valve and uses a donor valve in the pulmonary position which receives less stress than the aortic valve. The Ross procedure aims to improve valve durability with less clotting, avoiding use of blood thinners. Patients and physicians need a large, high-quality study comparing the Ross procedure and standard valve replacement to know if either approach is better.

The investigators will perform a 3-year feasibility study in seven sites, in Canada and abroad, to test the study design and ability to do a larger, conclusive study comparing the impact of the Ross procedure to standard valve replacement on survival without valve-related life-threatening complications. Patients will be randomized, like flipping a coin, to receive the Ross or standard valve surgery. The goals are 1) to evaluate if the investigators can recruit 6 patients per site per year, 2) to test if the assigned procedure is performed in over 90% of study patients, and 3) to see how many mechanical vs. tissue valves are used in the standard valve group. Patients eligible but not enrolled in the trial will be asked if the investigators can collect some data on how they do after their surgery. If the investigators show the study is feasible, they will proceed to the full study and will include the feasibility patients in the full study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years
2. Undergoing clinically indicated aortic valve replacement
3. Provided written informed consent

Exclusion Criteria:

1. Previous valve replacement not in the aortic position
2. Patients undergoing concomitant CABG or other valve procedure during aortic valve replacement
3. Known connective tissue disease
4. Severe (grade 3 or 4) right or left ventricular dysfunction
5. Pulmonary valve dysfunction or anomaly not compatible with the Ross procedure (as determined by the consulting cardiac surgeon)
6. Life expectancy less than 5 years (as determined by the consulting cardiac surgeon)
7. Documented severe aortic insufficiency not solely due to leaflet issue
8. Previous intervention on the pulmonary valve

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Full trial primary outcome - The rate of survival free of a composite of life-threatening valve-related complications (major bleeding, stroke or systemic thromboembolism, valve thrombosis, and operated-on valve reintervention) | Through trial completion, estimated to be 10 years
  The primary outcome is the rate of survival free of life-threatening valve-related complications (major bleeding, stroke or systemic thromboembolism, valve thrombosis, and operated-on valve reintervention) over duration of follow-up. Assessment of this composite over time is particularly important, as the Ross procedure may show initial benefit secondary to thromboembolic and bleeding reduction, however should the technique show high late rates of reoperation as suggested in some observational literature, the effect magnitude may change significantly over time.
Measure the pilot trial capacity to enrol a mean of 6 patients per centre per year to determine the feasibility of a full trial | Through completion of the pilot trial, estimated to be 3 years
  The outcome measures of the pilot trial, in order of importance, are:
  To evaluate the capacity to enroll a mean of 6 patients per centre per year.
The rate of compliance with allocation in the pilot trial to determine the feasibility of a full trial | Through completion of the pilot trial, estimated to be 3 years
  To determine the rate of compliance with randomization allocation.
Measure the proportions of type of conventional valve used in the pilot trial | Through completion of the pilot trial, estimated to be 3 years
  To validate the proportion of mechanical (at least 65%) versus biological (at most 35%) valves in the conventional arm.

SECONDARY OUTCOMES:
The rate of perioperative and non-perioperative major bleeding over the duration of patient follow-up | Through trial completion, estimated to be 10 years
  Perioperative (index surgery only) Intraoperative: After administration of protamine, delay of chest closure for bleeding > 500 mL/hr requiring packing and transfusion of more than 3 units red blood cells /whole blood.
  Upon leaving OR to 48hrs postop (modified BARC type 4)
  1. Intracranial bleeding within 48hrs
  2. Reoperation after sternum closure for purpose of controlling bleeding or relief of tamponade
  3. Transfusion of ≥ 5 units packed red blood cells /whole blood in the 48hr period
  4. Chest tube output ≥ 2L in the first 24hr
  Non-perioperative Per the International Society of Thrombosis and Hemostasis (ISTH) major bleeding definition.
The rate of stroke or systemic thromboembolism over the duration of patient follow-up | Through trial completion, estimated to be 10 years
  Stroke is acute focal brain dysfunction due to a vascular cause lasting ≥ 24 hrs in the absence of brain imaging or requires evidence of acute stroke on brain imaging (if there is a stroke documented by CT or MRI or at autopsy, the duration of symptoms/signs may be < 24 hours). Stroke is divided into 3 types: ischemic stroke, hemorrhagic stroke, and undetermined stroke. If death occurs within 24 hours, the neurological deficit must persist up to the time of death.
  Systemic arterial embolism is an abrupt vascular insufficiency associated with evidence of arterial occlusion in the absence of other likely mechanisms. Clinical signs/symptoms must be consistent with embolic arterial occlusion, there must be clear evidence of abrupt occlusion of a systemic artery, with at least one type of supporting evidence (surgical report indicating evidence of arterial embolism, pathological specimens related to embolism removal, imaging evidence consistent with arterial embolism, or autopsy report).
The rate of valve thrombosis per VARC criteria over the duration of patient follow-up | Through trial completion, estimated to be 10 years
  Valve thrombosis is defined as any thrombus not caused by infection attached to or near an operated valve that occludes part of the blood flow path, interferes with valve function, or is large enough to warrant treatment. Valve thrombus found at autopsy in a patient whose cause of death was not valve related or found at operation for and unrelated indication is to be counted as valve thrombosis.
The rate of operated-on valve reintervention over the duration of patient follow-up | Through trial completion, estimated to be 10 years
  Rate of valve reintervention Any surgical or percutaneous procedure that repairs, or otherwise alters or adjusts, or replaces a previously implanted prosthesis or valve.
Rate of mortality within 30 days post-operatively | 30 days
  Rate of mortality within 30 days post-operatively
Measure health related quality of life using the 36-Item Short Form Survey (SF-36) questionnaire over the duration of patient follow-up | Annually through trial completion, estimated to be 10 years
  The SF-36 is a health related quality of life questionnaire that measure eight health domains and each survey provides psychometrically-based physical component summary (PCS) and mental component summary (MCS) scores. The domains are physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. The questionnaire is calibrated such that scored values of 50 represent the norm and higher scored values according to the scoring key represent a more favourable health state. A baseline score will be obtained prior to the patient's surgery and the SF-36 will be administered annually thereafter over the duration of patient follow-up.
The rate of operated-valve endocarditis over the duration of patient follow-up | Through trial completion, estimated to be 10 years
  Defined as any infection involving a valve on which an operation has been performed. The diagnosis is based on one or more of the following: 1) reoperation with evidence of abscess, paravalvular leak, pus, or vegetation confirmed as secondary to infection by histologic or bacteriologic studies; 2) autopsy findings of abscess, pus, or vegetation involving an operated-on valve; or 3) the meeting of Duke criteria for endocarditis.
The rate of aortic valve re-intervention over the duration of patient follow-up | Through trial completion, estimated to be 10 years
  Any surgical or percutaneous procedure that repairs, or otherwise alters or adjusts, or replaces a previously implanted prosthesis or valve in the aortic position.
The rate of pulmonary valve re-intervention over the duration of patient follow-up | Through trial completion, estimated to be 10 years
  Any surgical or percutaneous procedure that repairs, or otherwise alters or adjusts, or replaces a previously implanted prosthesis or valve in the pulmonary position.
Mean aortic valve gradient | Through trial completion, estimated to be 10 years
  Measured through echocardiography
Mean pulmonic valve gradient | Through trial completion, estimated to be 10 years
  Measured through echocardiography
Severity of aortic valve regurgitation | Through trial completion, estimated to be 10 years
  Measured through echocardiography, categorized as mild, moderate, or severe
Severity of pulmonic valve regurgitation | Through trial completion, estimated to be 10 years
  Measured through echocardiography, categorized as mild, moderate, or severe

OTHER OUTCOMES:
Rate of myocardial infarction | 30 days postoperatively
  Myocardial infarction (Fourth universal definition)
  Occurring after 48 hrs post-operative, clinical evidence of acute myocardial injury with detection of a rise and/or fall of cTn values with at least one value above the 99th percentile URL and at least one of:
  * Symptoms of myocardial ischemia
  * New ischemic ECG changes
  * Development of pathological Q waves
  * Imaging evidence of new loss of viable myocardium or a new regional wall motion abnormality in a pattern consistent with an ischemic etiology; indication of a coronary thrombus by angiography or autopsy.
Rate of acute renal failure by Acute Kidney Injury Network classification | 30 days postoperatively
  Acute renal failure By AKIN classification - An abrupt (within 48 hours) reduction in kidney function currently defined as an absolute increase in serum creatinine of more than or equal to 0.3 mg/dl (≥ 26.4 μmol/l), a percentage increase in serum creatinine of more than or equal to 50% (1.5-fold from baseline), or a reduction in urine output (documented oliguria of less than 0.5 ml/kg per hour for more than six hours).
Rate of need for acute renal replacement therapy | 30 days postoperatively
  The rate of patients requiring new renal replacement therapy within 30 days of surgery.
Rate of surgical re-exploration of the mediastinum for bleeding | 30 days postoperatively
  Surgical re-exploration of the mediastinum for bleeding
Rate of deep mediastinal wound infection | 30 days postoperatively
  Deep mediastinal wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Richard Whitlock, MD, PhD, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Whitlock R, Belley-Cote E, Rega F, Chu MWA, McClure GR, Hronyecz H, Verbrugghe P, Devereaux PJ, Bangdiwala S, Eikelboom J, Brady K, Sharifulin R, Bogachev-Prokophiev A, Stoica S. Ross for Valve replacement In AduLts (REVIVAL) pilot trial: rationale and design of a randomised controlled trial. BMJ Open. 2021 Sep 16;11(9):e046198. doi: 10.1136/bmjopen-2020-046198. PMID 34531204